CLINICAL TRIAL: NCT00652002
Title: A 12 Week, Randomized, Double-blind, Double-dummy, Placebo-controlled Trial of Symbicort TM (160/4.5mcg) Versus Its Mono-products (Budesonide and Formoterol) in Adolescents (at Least 12 Years of Age) and Adults With Asthma - SPRUCE 160/4.5
Brief Title: Efficacy of Symbicort Versus Its Monocomponents - SPRUCE 160/4.5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SD-039-0717; D5896C00717
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; Symbicort; budesonide/formoterol; budesonide; formoterol
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: budesonide/formoterol
- 2 (Active Comparator): budesonide
  Interventions: Drug: budesonide
- 3 (Active Comparator): formoterol
  Interventions: Drug: formoterol

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
  Arms: 1
Drug: budesonide
  Arms: 2
Drug: formoterol
  Arms: 3

SUMMARY:
The purpose of this study is to compare Symbicort with budesonide alone and with formoterol alone in the treatment of asthma in adolescents and adults

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age
* Diagnosis of asthma
* Baseline lung function test results as determined by protocol and required and received treatment with inhaled corticosteroids and/or lung treatments specified in protocol within the timeframe and doses specified in the protocol

Exclusion Criteria:

* Has required treatment with non-inhaled corticosteroids within previous 4 weeks, has sensitivity to drugs specified in the protocol or requires treatment with beta-blockers
* Had cancer within previous 5 years or currently has any other significant disease or disorder as judged by the investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2002-07; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
12 hour serial FEV1 measurements and withdrawals due to asthma exacerbation | FEV1: before start of tretment and at 2 and 12 weeks after start of treatment. Withdrawals: throughout the treatment period

SECONDARY OUTCOMES:
Lung function, asthma symptoms, use of rescue medication, adverse events and other safety assessments | Throughout the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca

REFERENCES:
- [Derived] Tashkin DP, Moore GE, Trudo F, DePietro M, Chipps BE. Assessment of Consistency of Fixed Airflow Obstruction Status during Budesonide/Formoterol Treatment and Its Effects on Treatment Outcomes in Patients with Asthma. J Allergy Clin Immunol Pract. 2016 Jul-Aug;4(4):705-12. doi: 10.1016/j.jaip.2016.02.014. Epub 2016 Mar 30. PMID 27039236
- [Derived] Tashkin DP, Chipps BE, Trudo F, Zangrilli JG. Fixed airflow obstruction in asthma: a descriptive study of patient profiles and effect on treatment responses. J Asthma. 2014 Aug;51(6):603-9. doi: 10.3109/02770903.2014.895012. Epub 2014 Mar 19. PMID 24524222
- [Derived] Murphy KR, Uryniak T, Martin UJ, Zangrilli J. The effect of budesonide/formoterol pressurized metered-dose inhaler on predefined criteria for worsening asthma in four different patient populations with asthma. Drugs R D. 2012 Mar 1;12(1):9-14. doi: 10.2165/11630600-000000000-00000. PMID 22329608